CLINICAL TRIAL: NCT03692871
Title: A Phase 3, Multicenter, Randomized, Double-blind, Active Comparator-controlled Study to Evaluate the Safety and Tolerability of V114 in Healthy Infants (PNEU-LINK)
Brief Title: A Study to Evaluate the Safety and Tolerability of V114 and Prevnar 13™ in Healthy Infants (V114-031/PNEU-LINK)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: V114-031; V114-031 (Other: Merck); 2018-003308-38 (EudraCT Number)
Record Dates: First submitted 2018-09-28; First posted 2018-10-02 (Actual); Results first posted 2022-05-10 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Pneumococcal Infections
MeSH Terms: conditions — Pneumococcal Infections | interventions — 13-valent pneumococcal vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- V114 (Experimental): Participants will receive a single 0.5 mL intramuscular (IM) injection of V114 at approximately 2 months of age (Vaccination 1); approximately 4 months of age (Vaccination 2); approximately 6 months of age (Vaccination 3); and approximately 12-15 months of age (Vaccination 4).
  Interventions: Biological: V114
- Prevnar 13™ (Active Comparator): Participants will receive a single 0.5 mL IM injection of Prevnar 13™ at approximately 2 months of age (Vaccination 1); approximately 4 months of age (Vaccination 2); approximately 6 months of age (Vaccination 3); and approximately 12-15 months of age (Vaccination 4).
  Interventions: Biological: Prevnar 13™

INTERVENTIONS:
Biological: V114 — V114 pneumococcal capsular polysaccharide serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 22F, 23F, 33F (2 mcg each), and serotype 6B (4 mcg) in each 0.5 mL dose
  Other Names: VAXNEUVANCE™; Pneumococcal 15-Valent Conjugate Vaccine
  Arms: V114
Biological: Prevnar 13™ — Prevnar 13™ pneumococcal capsular polysaccharide serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 23F (2.2 mcg each) and 6B (4.4 mcg) in each 0.5 ml dose
  Arms: Prevnar 13™

SUMMARY:
This study is designed to evaluate the safety and tolerability of V114 and Prevnar 13™ in healthy infants. This study will include both full-term infants (≥37 weeks gestational age) and premature infants (<37 weeks gestational age). Premature infants will be included in a Premature Infant Immunogenicity Substudy, which will assess immunogenicity and safety following administration of V114 or Prevnar 13™.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (based on a review of medical history and physical examination) based on the clinical judgment of the investigator
* Male or female approximately 2 months of age, from 42 days to 90 days inclusive, at the time of obtaining the informed consent
* Have a legally acceptable representative who understands the study procedures, alternate treatments available, and risks involved with the study and voluntarily agrees to participate by giving written informed consent.

Exclusion Criteria:

* History of Invasive Pneumococcal Disease (IPD) (positive blood culture, positive cerebrospinal fluid culture, or other sterile site) or known history of other culture positive pneumococcal disease
* Known hypersensitivity to any component of the pneumococcal conjugate vaccine (PCV) or any diphtheria toxoid containing vaccine
* Known or suspected impairment of immunological function
* History of congenital or acquired immunodeficiency
* Has or his/her mother has a documented human immunodeficiency virus (HIV) infection
* Known or history of functional or anatomic asplenia
* Failure to thrive based on the clinical judgment of the investigator
* Known coagulation disorder contraindicating intramuscular vaccination
* History of autoimmune disease (including but not limited to systemic lupus erythematosus, antiphospholipid syndrome, Behcet's disease, autoimmune thyroid disease, polymyositis and dermatomyositis, scleroderma, type 1 diabetes mellitus, or other autoimmune disorders)
* Known neurologic or cognitive behavioral disorder, including encephalitis/myelitis, acute disseminating encephalomyelitis, pervasive development disorder, and related disorders
* Received a dose of any pneumococcal vaccine prior to study entry
* Received a blood transfusion or blood products, including immunoglobulins, before receipt of first dose of study vaccine
* Participated in another clinical study of an investigational product before the beginning or anytime during the duration of the current clinical study. Participants enrolled in observational studies may be included.
* Has any other reason that, in the opinion of the investigator, may interfere with the evaluation required by the study
* Has an immediate family member who is investigational site or Sponsor staff directly involved with this study.

Ages: 42 Days to 90 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2409 (Actual)
Dates: Start 2018-12-14 (Actual); Primary Completion 2021-03-26 (Actual); Study Completion 2021-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (76):
- United States (22):
  - Premier Health Research Center, LLC ( Site 0005), Downey, California
  - Beach Pediatrics ( Site 0040), Huntington Beach, California
  - Khruz Biotechnology Research Institute ( Site 0006), San Diego, California
  - Kaiser Permanente - San Jose ( Site 0036), San Jose, California
  - Kaiser Permanente - Santa Clara ( Site 0027), Santa Clara, California
  - Children's Research, LLC ( Site 0025), Lake Mary, Florida
  - Advanced Research For Health Improvement LLC ( Site 0030), Naples, Florida
  - Pediatric Partners, P.A. ( Site 0010), Overland Park, Kansas
  - Novak Center for Childrens Health ( Site 0033), Louisville, Kentucky
  - Medpharmics, LLC ( Site 0037), Metairie, Louisiana
  - Child Health Care Associates ( Site 0024), East Syracuse, New York
  - Primedical Clinical Research ( Site 0035), Dayton, Ohio
  - Allegheny Health & Wellness Pavilion West ( Site 0034), Erie, Pennsylvania
  - CCP- Kid's Way ( Site 0008), Hermitage, Pennsylvania
  - Thomas Jefferson University ( Site 0029), Philadelphia, Pennsylvania
  - Medical Research South, LLC ( Site 0013), Charleston, South Carolina
  - Pediatric Associates [Houston, TX] ( Site 0039), Houston, Texas
  - University of Texas Medical Branch ( Site 0018), League City, Texas
  - Tanner Clinic ( Site 0009), Layton, Utah
  - Wee Care Pediatrics ( Site 0031), Layton, Utah
  - Wee Care Pediatrics ( Site 0020), Roy, Utah
  - University of Wisconsin American Family Children's Hospital ( Site 0023), Madison, Wisconsin
- Australia (3):
  - Monash Children s Hospital ( Site 0093), Clayton, Victoria
  - Perth Children s Hospital ( Site 0092), Nedlands
  - Children, Youth and Woman's Health Service ( Site 0094), North Adelaide
- Canada (8):
  - Alberta Children s Hospital ( Site 0048), Calgary, Alberta
  - Vaccine Evaluation Center BC Children s Hospital Research Institute ( Site 0046), Vancouver, British Columbia
  - IWK Health Centre [Halifax, Canada] ( Site 0043), Halifax, Nova Scotia
  - Medicor Research Inc. ( Site 0041), Greater Sudbury, Ontario
  - Hamilton Medical Research Group ( Site 0049), Hamilton, Ontario
  - CHU Sainte Justine ( Site 0047), Montreal, Quebec
  - McGill University Health Centre - Vaccine Study Centre ( Site 0045), Pierrefonds, Quebec
  - CHUQ - Unite de Recherche en Sante Publique ( Site 0042), Québec, Quebec
- Finland (10):
  - Espoon rokotetutkimuskeskus ( Site 0066), Espoo
  - Tampereen yliopisto Etela-Helsingin Rokotetutkimusklinikka ( Site 0064), Helsinki
  - Ita-Helsingin Rokotetutkimuskeskus ( Site 0065), Helsinki
  - Jarvenpaan rokotetutkimuskeskus ( Site 0067), Jarvenpaa
  - Kokkolan rokotetutkimusklinikka ( Site 0071), Kokkola
  - Tampereen yliopisto Oulun rokotetutkimusklinikka ( Site 0072), Oulu
  - Porin Rokotetutkimusklinikka ( Site 0069), Pori
  - Seinajoki Vaccine Research Center ( Site 0070), Seinäjoki
  - Tampereen yliopisto - Tampereen rokotetutkimusklinikka ( Site 0063), Tampere
  - Turun rokotetutkimuskeskus ( Site 0068), Turku
- Germany (9):
  - Kinderarztpraxis ( Site 0124), Aschaffenburg
  - Kinderarztpraxis ( Site 0123), Bramsche
  - Kinderarztpraxis Dr. Friedrich Kaiser & Dr. Marinesse ( Site 0085), Hamburg
  - Kinderarztpraxis ( Site 0081), Hürth
  - Kinderarztpraxis Dr. Muehlschlegel - Dr. Goetz ( Site 0122), Lauffen am Neckar
  - Kinderarztpraxis ( Site 0080), Mönchengladbach
  - Kinderarztpraxis Matthias Donner Dr. M. Luechtrath ( Site 0091), Munchengladbach
  - Kinderarztpraxis ( Site 0084), Schönau
  - Kinderaerztliche Gemeinschaftspraxis Drs. Westerholt/Matyas ( Site 0083), Wolfsburg
- Israel (7):
  - Soroka University Medical Center ( Site 0077), Beersheba
  - Soroka University Medical Center - Ramot Family health center ( Site 0078), Beersheba
  - Rambam Medical Center ( Site 0076), Haifa
  - Rambam Medical Center- Keriat Eliezer Family Health Center ( Site 0138), Haifa
  - Rambam Medical Center- Neve David Family Health Center ( Site 0139), Haifa
  - Soroka Medical Center_ Hura Family health center ( Site 0137), Hura
  - Soroka University Medical Center - Rahat Family health center ( Site 0079), Rahat
- Malaysia (5):
  - Klinik Kesihatan Greentown ( Site 0132), Ipoh, Perak
  - Sarawak General Hospital ( Site 0107), Kuching, Sarawak
  - Hospital Sibu ( Site 0111), Sibu, Sarawak
  - Universiti Malaya Medical Center-Clinical Investigation Center ( Site 0108), Kuala Lumpur
  - Klinik Kesihatan Pandamaran ( Site 0110), Port Klang
- Peru (3):
  - Hospital Nacional Docente Madre - Nino San Bartolome ( Site 0057), Lima
  - Instituto de Investigacion Nutricional ( Site 0058), Lima
  - Clinica Peruano Americana S.A. ( Site 0061), Trujillo
- Taiwan (4):
  - Taichung Veterans General Hospital ( Site 0100), Taichung
  - National Taiwan University Hospital ( Site 0097), Taipei
  - Mackay Memorial Hospital ( Site 0099), Taipei
  - Chang Gung Medical Foundation. Linkou ( Site 0098), Taoyuan District
- Thailand (5):
  - Chulalongkorn University ( Site 0102), Bangkok
  - Siriraj Hospital ( Site 0101), Bangkok
  - Maharaj Nakorn Chiang Mai Hospital ( Site 0103), Chiang Mai
  - Prince of Songkla University, Faculty of Medicine ( Site 0105), Hat Yai
  - Srinagarind Hospital. Khon Kaen University ( Site 0104), Khon Kaen

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Banniettis N, Horn M, Sadarangani M, Patel SM, Greenberg D, Oberdorfer P, Klein NP, Rupp R, Dagan R, Richmond P, Lumley J, Zhou W, Shi Y, Tamms G, Feemster K, Lupinacci R, Musey L, Bickham K; V114-031 (PNEU-LINK) study group. Safety and Tolerability of V114 Pneumococcal Vaccine in Infants: A Phase 3 Study. Pediatrics. 2023 Jul 1;152(1):e2022060428. doi: 10.1542/peds.2022-060428. PMID 37309607

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study enrolled healthy infants. Other inclusion criteria applied.
Groups:
- V114: Participants received a single 0.5 mL intramuscular (IM) injection of V114 at approximately 2 months of age (Vaccination 1); approximately 4 months of age (Vaccination 2); approximately 6 months of age (Vaccination 3); and approximately 12-15 months of age (Vaccination 4).
- Prevnar 13™: Participants received a single 0.5 mL IM injection of Prevnar 13™ at approximately 2 months of age (Vaccination 1); approximately 4 months of age (Vaccination 2); approximately 6 months of age (Vaccination 3); and approximately 12-15 months of age (Vaccination 4).
Period: Overall Study
Arm/Group | V114 | Prevnar 13™
Started | 1972 | 437
Completed | 1847 | 400
Not Completed | 125 | 37
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 24 | 9
Not completed — Physician Decision | 22 | 7
Not completed — Protocol Deviation | 1 | 0
Not completed — Withdrawal by Parent/Guardian | 77 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | V114 | Prevnar 13™ | Total
Number analyzed (Participants) | 1972 | 437 | 2409
Age, Continuous [Mean (Standard Deviation); unit: weeks] | 8.7 (1.5) | 8.8 (1.5) | 8.7 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 948 | 227 | 1175
  Male | 1024 | 210 | 1234
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 293 | 74 | 367
  Not Hispanic or Latino | 1678 | 362 | 2040
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 64 | 20 | 84
  Asian | 730 | 152 | 882
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 54 | 19 | 73
  White | 966 | 214 | 1180
  More than one race | 154 | 31 | 185
  Unknown or Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Solicited Injection-site Adverse Event
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. Solicited injection-site AEs included injection-site erythema (redness), injection-site induration (hard lump), injection-site pain (tenderness), and injection-site swelling.
Time Frame: Up to Day 14 after each study vaccination
Population: All randomized participants who received at least 1 dose of study vaccination
Measure: Number; unit: Percentage of participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 1965 | 433
Percentage of participants
  Injection-site erythema | 43.9 | 36.0
  Injection-site induration | 25.3 | 25.6
  Injection-site pain | 42.9 | 36.5
  Injection-site swelling | 27.9 | 23.3
Statistical Analysis 1: Comparison: V114 vs Prevnar 13™; Injection-site erythema; Test type: Other; p = 0.003, Miettinen & Nurminen method; Difference in Percentage = 7.9, 95% CI 2-sided [2.8 to 12.8]
Statistical Analysis 2: Comparison: V114 vs Prevnar 13™; Injection-site induration; Test type: Other; p = 0.882, Miettinen & Nurminen method; Difference in Percentage = -0.3, 95% CI 2-sided [-5.0 to 4.0]
Statistical Analysis 3: Comparison: V114 vs Prevnar 13™; Injection-site pain; Test type: Other; p = 0.014, Miettinen & Nurminen method; Difference in Percentage = 6.4, 95% CI 2-sided [1.3 to 11.3]
Statistical Analysis 4: Comparison: V114 vs Prevnar 13™; Injection-site swelling; Test type: Other; p = 0.051, Miettinen & Nurminen method; Difference in Percentage = 4.6, 95% CI 2-sided [0.0 to 8.9]

2. Primary Outcome: Percentage of Participants With a Solicited Systemic Adverse Event
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. Solicited systemic AEs included decreased appetite, irritability, somnolence (drowsiness), and urticaria (hives or welts).
Time Frame: Up to Day 14 after each study vaccination
Population: All randomized participants who received at least 1 dose of study vaccination
Measure: Number; unit: Percentage of participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 1965 | 433
Percentage of participants
  Decreased appetite | 41.6 | 36.0
  Irritability | 74.9 | 69.3
  Somnolence | 55.4 | 55.0
  Urticaria | 5.9 | 6.7
Statistical Analysis 1: Comparison: V114 vs Prevnar 13™; Decreased appetite; Test type: Other; p = 0.033, Miettinen & Nurminen method; Difference in Percentage = 5.5, 95% CI 2-sided [0.4 to 10.5]
Statistical Analysis 2: Comparison: V114 vs Prevnar 13™; Irritability; Test type: Other; p = 0.016, Miettinen & Nurminen method; Difference in Percentage = 5.6, 95% CI 2-sided [1.0 to 10.5]
Statistical Analysis 3: Comparison: V114 vs Prevnar 13™; Somnolence; Test type: Other; p = 0.878, Miettinen & Nurminen method; Difference in Percentage = 0.4, 95% CI 2-sided [-4.7 to 5.6]
Statistical Analysis 4: Comparison: V114 vs Prevnar 13™; Urticaria; Test type: Other; p = 0.503, Miettinen & Nurminen method; Difference in Percentage = -0.8, 95% CI 2-sided [-3.8 to 1.5]

3. Primary Outcome: Percentage of Participants With a Vaccine-related Serious Adverse Event
Description: A serious adverse event (SAE) is an AE that results in death, is life-threatening, requires or prolongs an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, or is another important medical event deemed such by medical or scientific judgment. SAEs that were reported by the investigator to be at least possibly related to the study vaccination were summarized.
Time Frame: Up to 6 months after Vaccination 4 (up to 19 months after Vaccination 1)
Population: All randomized participants who received at least 1 dose of study vaccination
Measure: Number; unit: Percentage of participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 1965 | 433
Percentage of participants | 0.1 | 0
Statistical Analysis 1: Comparison: V114 vs Prevnar 13™; Percentage of participants with a vaccine-related SAE; Test type: Other; Difference in Percentage = 0.1, 95% CI 2-sided [-0.8 to 0.4]

4. Secondary Outcome: Geometric Mean Concentration (GMC) of Serotype-specific Immunoglobulin G (IgG) at 30 Days After Vaccination 3 (Premature Infants Only)
Description: The GMC of IgG serotype-specific antibodies to the 13 serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) included in V114 and Prevnar 13™ and 2 serotypes (22F and 33F) unique to V114 were quantitated from participants' sera by a multiplex electrochemiluminescence (ECL) assay. This endpoint was part of a Premature Infant Immunogenicity Substudy.
Time Frame: 30 days after Vaccination 3 (approximately 5 months after Vaccination 1)
Population: All randomized participants in the Premature Infant Immunogenicity Substudy who did not have protocol deviations that could have substantially affected the results of the immunogenicity analysis and who had sufficient data to perform the analysis for each serotype
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 38 | 35
μg/mL
  Serotype 1 | 1.15 [0.88 to 1.52] | 1.61 [1.25 to 2.09]
  Serotype 3 | 0.86 [0.65 to 1.13] | 0.58 [0.45 to 0.76]
  Serotype 4 | 1.41 [1.01 to 1.99] | 1.27 [0.96 to 1.68]
  Serotype 5 | 1.48 [1.04 to 2.10] | 1.66 [1.09 to 2.53]
  Serotype 6A | 1.37 [0.95 to 1.96] | 3.19 [2.31 to 4.43]
  Serotype 6B | 1.69 [1.15 to 2.48] | 2.53 [1.64 to 3.89]
  Serotype 7F | 1.95 [1.46 to 2.62] | 2.92 [2.21 to 3.87]
  Serotype 9V | 1.47 [1.08 to 2.00] | 1.50 [1.07 to 2.12]
  Serotype 14 | 4.38 [3.18 to 6.03] | 6.52 [4.35 to 9.77]
  Serotype 18C | 1.46 [1.08 to 1.96] | 1.54 [1.16 to 2.04]
  Serotype 19A | 1.63 [1.25 to 2.13] | 3.00 [2.18 to 4.11]
  Serotype 19F | 2.03 [1.53 to 2.68] | 2.78 [2.17 to 3.58]
  Serotype 23F | 1.17 [0.81 to 1.70] | 1.18 [0.82 to 1.68]
  Serotype 22F | 4.33 [3.18 to 5.90] | 0.05 [0.03 to 0.07]
  Serotype 33F | 1.58 [0.93 to 2.69] | 0.05 [0.04 to 0.08]

5. Secondary Outcome: GMC of Serotype-specific IgG Before Vaccination 4 (Premature Infants Only)
Description: as for outcome 4
Time Frame: Before Vaccination 4 (10-13 months after Vaccination 1)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 38 | 40
μg/mL
  Serotype 1 | 0.30 [0.24 to 0.38] | 0.47 [0.38 to 0.59]
  Serotype 3 | 0.22 [0.16 to 0.29] | 0.13 [0.10 to 0.17]
  Serotype 4 | 0.24 [0.19 to 0.31] | 0.31 [0.24 to 0.38]
  Serotype 5 | 0.77 [0.60 to 1.01] | 0.89 [0.65 to 1.22]
  Serotype 6A | 0.32 [0.24 to 0.43] | 0.72 [0.52 to 0.99]
  Serotype 6B | 0.59 [0.47 to 0.75] | 0.61 [0.43 to 0.87]
  Serotype 7F | 0.57 [0.44 to 0.73] | 0.95 [0.74 to 1.21]
  Serotype 9V | 0.40 [0.32 to 0.51] | 0.46 [0.35 to 0.62]
  Serotype 14 | 1.14 [0.84 to 1.54] | 2.22 [1.73 to 2.84]
  Serotype 18C | 0.35 [0.28 to 0.45] | 0.36 [0.27 to 0.49]
  Serotype 19A | 0.38 [0.29 to 0.51] | 0.81 [0.52 to 1.24]
  Serotype 19F | 0.41 [0.31 to 0.53] | 0.69 [0.52 to 0.90]
  Serotype 23F | 0.33 [0.24 to 0.45] | 0.37 [0.26 to 0.52]
  Serotype 22F | 1.24 [0.98 to 1.58] | 0.05 [0.04 to 0.07]
  Serotype 33F | 1.09 [0.82 to 1.45] | 0.05 [0.04 to 0.07]

6. Secondary Outcome: GMC of Serotype-specific IgG at 30 Days After Vaccination 4 (Premature Infants Only)
Description: as for outcome 4
Time Frame: 30 days after Vaccination 4 (11-14 months after Vaccination 1)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 34 | 39
μg/mL
  Serotype 1 | 1.56 [1.19 to 2.06] | 1.96 [1.54 to 2.50]
  Serotype 3 | 1.04 [0.80 to 1.36] | 0.79 [0.60 to 1.06]
  Serotype 4 | 1.55 [1.11 to 2.16] | 1.61 [1.21 to 2.15]
  Serotype 5 | 3.30 [2.34 to 4.65] | 3.60 [2.53 to 5.13]
  Serotype 6A | 4.18 [3.17 to 5.49] | 6.38 [4.69 to 8.68]
  Serotype 6B | 6.62 [5.24 to 8.37] | 6.75 [4.43 to 10.28]
  Serotype 7F | 4.01 [2.98 to 5.40] | 5.10 [3.76 to 6.90]
  Serotype 9V | 3.10 [2.36 to 4.08] | 3.09 [2.31 to 4.12]
  Serotype 14 | 5.40 [3.89 to 7.49] | 7.15 [5.33 to 9.61]
  Serotype 18C | 3.21 [2.32 to 4.45] | 2.77 [1.99 to 3.85]
  Serotype 19A | 4.96 [3.85 to 6.39] | 6.47 [4.46 to 9.40]
  Serotype 19F | 4.48 [3.51 to 5.73] | 4.83 [3.66 to 6.38]
  Serotype 23F | 2.38 [1.76 to 3.20] | 3.04 [2.16 to 4.27]
  Serotype 22F: number analyzed (Participants) | 34 | 38
  Serotype 22F | 9.83 [7.47 to 12.92] | 0.08 [0.07 to 0.11]
  Serotype 33F: number analyzed (Participants) | 34 | 37
  Serotype 33F | 5.46 [4.29 to 6.96] | 0.10 [0.07 to 0.13]

7. Secondary Outcome: Percentage of Participants Meeting Serotype-specific IgG Threshold of ≥0.35 μg/mL 30 Days After Vaccination 3 (Premature Infants Only)
Description: The GMC of IgG serotype-specific antibodies to the 13 serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) included in V114 and Prevnar 13™ and 2 serotypes (22F and 33F) unique to V114 were quantitated from participants' sera by a multiplex electrochemiluminescence (ECL) assay. Immunoglobulin G for the 15 serotypes contained in V114 vaccine was determined using a pneumococcal electrochemiluminescence (PnECL) assay. This endpoint was part of a Premature Infant Immunogenicity Substudy.
Time Frame: 30 days after Vaccination 3 (approximately 5 months after Vaccination 1)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 38 | 35
Percentage of participants
  Serotype 1 | 97.4 [86.2 to 99.9] | 97.1 [85.1 to 99.9]
  Serotype 3 | 89.5 [75.2 to 97.1] | 74.3 [56.7 to 87.5]
  Serotype 4 | 94.7 [82.3 to 99.4] | 97.1 [85.1 to 99.9]
  Serotype 5 | 97.4 [86.2 to 99.9] | 88.6 [73.3 to 96.8]
  Serotype 6A | 97.4 [86.2 to 99.9] | 97.1 [85.1 to 99.9]
  Serotype 6B | 92.1 [78.6 to 98.3] | 94.3 [80.8 to 99.3]
  Serotype 7F | 97.4 [86.2 to 99.9] | 100 [90.0 to 100.0]
  Serotype 9V | 97.4 [86.2 to 99.9] | 94.3 [80.8 to 99.3]
  Serotype 14 | 100 [90.7 to 100.0] | 97.1 [85.1 to 99.9]
  Serotype 18C | 97.4 [86.2 to 99.9] | 94.3 [80.8 to 99.3]
  Serotype 19A | 94.7 [82.3 to 99.4] | 97.1 [85.1 to 99.9]
  Serotype 19F | 97.4 [86.2 to 99.9] | 100 [90.0 to 100.0]
  Serotype 23F | 89.5 [75.2 to 97.1] | 94.3 [80.8 to 99.3]
  Serotype 22F | 97.4 [86.2 to 99.9] | 2.9 [0.1 to 14.9]
  Serotype 33F | 86.8 [71.9 to 95.6] | 2.9 [0.1 to 14.9]

ADVERSE EVENTS:
Time Frame: Non-serious AEs: up to 14 days after each vaccination dose; serious AEs and deaths (all causes): up to 6 months after Vaccination 4 (up to 19 months after Vaccination 1)
Description: The safety analysis population included all randomized participants who received at least 1 dose of study vaccination.
  The analysis population for All-Cause Mortality included all randomized participants.
Arm/Group | V114 | Prevnar 13™
All-Cause Mortality (participants affected / at risk) | 1/1972 | 1/437
Serious Adverse Events (participants affected / at risk) | 192/1965 | 45/433
Other Adverse Events (participants affected / at risk) | 1807/1965 | 395/433
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V114 (N=1965) | Prevnar 13™ (N=433)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Congenital absence of bile ducts (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 8 (8) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 27 (29) | 7 (10)
Bronchitis (Infections and infestations) | 8 (8) | 2 (2)
Bronchitis viral (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Coxsackie viral infection (Infections and infestations) | 1 (1) | 0 (0)
Croup infectious (Infections and infestations) | 2 (2) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 3 (3) | 0 (0)
Enterovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Escherichia pyelonephritis (Infections and infestations) | 8 (8) | 1 (1)
Escherichia sepsis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 6 (6) | 1 (1)
Exanthema subitum (Infections and infestations) | 7 (7) | 1 (1)
Gastroenteritis (Infections and infestations) | 15 (17) | 0 (0)
Gastroenteritis adenovirus (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis norovirus (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis salmonella (Infections and infestations) | 4 (4) | 0 (0)
Gastroenteritis shigella (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 5 (5) | 1 (1)
Hand-foot-and-mouth disease (Infections and infestations) | 3 (3) | 0 (0)
Herpangina (Infections and infestations) | 3 (3) | 1 (1)
Influenza (Infections and infestations) | 4 (4) | 3 (3)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Mastoiditis (Infections and infestations) | 1 (1) | 0 (0)
Metapneumovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 1 (1)
Pertussis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 12 (13) | 4 (4)
Pneumonia influenzal (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia parainfluenzae viral (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia respiratory syncytial viral (Infections and infestations) | 5 (5) | 2 (2)
Pneumonia viral (Infections and infestations) | 7 (7) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Rectal abscess (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 9 (10) | 4 (4)
Respiratory syncytial virus bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 2 (2) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 3 (3) | 0 (0)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 2 (3) | 1 (1)
Urinary tract infection enterococcal (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 4 (4) | 0 (0)
Viral pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Accidental exposure to product (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chemical poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Chronic recurrent multifocal osteomyelitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Oligoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hepatoblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Febrile convulsion (Nervous system disorders) | 4 (4) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Myoclonus (Nervous system disorders) | 1 (1) | 0 (0)
Paroxysmal choreoathetosis (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V114 (N=1965) | Prevnar 13™ (N=433)
Diarrhoea (Gastrointestinal disorders) | 188 (235) | 40 (49)
Vomiting (Gastrointestinal disorders) | 116 (135) | 19 (20)
Injection site erythema (General disorders) | 863 (1528) | 156 (272)
Injection site induration (General disorders) | 497 (885) | 111 (205)
Injection site pain (General disorders) | 843 (1580) | 158 (288)
Injection site swelling (General disorders) | 549 (929) | 101 (163)
Pyrexia (General disorders) | 775 (1533) | 176 (329)
Nasopharyngitis (Infections and infestations) | 158 (182) | 37 (41)
Upper respiratory tract infection (Infections and infestations) | 129 (139) | 30 (32)
Decreased appetite (Metabolism and nutrition disorders) | 817 (1664) | 156 (302)
Somnolence (Nervous system disorders) | 1088 (2696) | 238 (590)
Irritability (Psychiatric disorders) | 1472 (5402) | 300 (1053)
Urticaria (Skin and subcutaneous tissue disorders) | 115 (139) | 29 (40)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigators agree to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-11): https://cdn.clinicaltrials.gov/large-docs/71/NCT03692871/Prot_SAP_000.pdf